CLINICAL TRIAL: NCT01224951
Title: Development and Validation of a Sputum Biomarker mRNA Panel for the Diagnostic Work-up of Asthma 2
Acronym: BioSput-Air
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dominque Bullens, prof. dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Biomarker sputum airway study2
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Qvar 100 (Active Comparator): Patients will be randomized to receive either the active arm (3/4) or a SABA as rescue medication (1/4). The patient will be asked to take Qvar 100 (2puffs) in the morning and in the evening.
  Daily dose (400 microgram).
  Interventions: Drug: Beclomethasone
- Control (No Intervention): Patients are allowed to use their SABA as rescue medication only. During the last 4 weeks, the patients will receive 400 microgram of Qvar.

INTERVENTIONS:
Drug: Beclomethasone — 400 microgram of beclomethasone will be given to the patients in arm 1. During the last 4 weeks, the patients will receive additional 400 microgram of Qvar.
  Other Names: Qvar 100
  Arms: Qvar 100

SUMMARY:
The main objectives of the study are:

-to unravel the importance of molecular phenotyping in predicting the response to classical anti-asthma treatment (inhaled corticosteroids)

The investigators have developed a non-invasive technique based on mRNA analysis of induced sputum that enables us to study airway inflammation in detail. This technique forms the basis for our current project based on the following hypotheses:

1. different molecular asthma phenotypes exist: a Th2 phenotype and a non Th2 phenotype as reported by Woodruff and colleagues (Woodruff PG et al). Sputum mRNA cytokine levels can be used to diagnose Th2 asthma and discriminate this from non-Th2 asthma.
2. Based on our previous research and preliminary data that non-Th2 asthma can be further divided in Th17 asthma and Th1+Th2 asthma; besides these, a fourth group without Th2, Th17 or Th1 characteristics also exist. The investigators hypothesize that the epithelial cell cytokine, TSLP, can be increased as an early marker of airway inflammation in this latter group.
3. these subgroups have different responses to anti-inflammatory treatment.

ELIGIBILITY:
Inclusion Criteria:

* steroid naive asthmatics

Exclusion Criteria:

* viral/bacterial/fungal infection +fever(<1month)
* asthma exacerbation (<3months)
* other airway diseases (CF, ciliary dyskinesia, bronchiectasis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-02 (Actual); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
sputum cytokine mRNA levels | 6 and 10 weeks

SECONDARY OUTCOMES:
steroid-responsiveness | 6 and 10 weeks
  We will evaluate steroid-responsiveness both by objective measurements (lung function parameters) and asthma scores

CONTACTS AND LOCATIONS:
Overall Officials: Dominique MA Bullens, MD, PhD, Principal Investigator — Lab of clinical immunology, O&N I Herestraat 49 - bus 811, 3000 Leuven, België; Sven F Seys, MSc, Study Director — Lab of clinical immunology, O&N I Herestraat 49 - bus 811, 3000 Leuven, België
Locations (1):
- University Hospital of Leuven, Leuven, Vlaams-Brabant, Belgium